## **Cover Page**

Official Title: Effect of Fan Therapy on Dyspnea Associated With Ticagrelor Administration

in Intensive Care Patients

**NCT Number:** Not yet assigned

Document Date: 18 July 2024

Prepared by: Emine Tuğba Yorulmaz, PhD Student

Supervised by: Asst. Prof. Arzu Erkoç

**Document Type**: Ethics Approval

## **Ethics Approval (İngilizce)**

Document Type: Study Protocol with SAP and/or ICF

Document Date: 18 July 2024

Subtitle: ATADEK Ethical Approval

### **Ethics Approval**

Reference Number: ATADEK-2024/10

Date: 18 July 2024

# **Principal Investigators:**

Dr. Öğr. Üyesi Arzu Erkoç

Arş. Gör. Emine Tuğba Yorulmaz

**Study Title:** Effect of Fan Therapy on Dyspnea Associated With Ticagrelor Administration in Intensive Care Patients

### **Approval Statement:**

The study protocol was reviewed at the ATADEK meeting on 18 July 2024 and approved with decision number 2024-10/449 as ethically acceptable for conduct according to medical ethical standards in Turkey.